CLINICAL TRIAL: NCT02377401
Title: A Randomized, Double Blinded, Parallel Study to Evaluate the Pharmacokinetics of Zanamivir After Single and Repeated Dose (300 mg and 600 mg) Infusion Administration in Healthy Chinese Adults
Brief Title: Pharmacokinetics of Zanamivir After Single and Repeated Dose Infusion Administration in Healthy Chinese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 117104
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Influenza, Human
Keywords: healthy volunteer; Zanamivir; pharmacokinetics; intravenous
MeSH Terms: conditions — Influenza, Human | interventions — Zanamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zanamivir 300 mg (Experimental): Subjects will receive a single dose of IV zanamivir 300 mg on Day 1 morning. The repeat dose session will begin on Day 3 evening. Subjects will receive IV zanamivir 300 mg every 12 hours for 5 days. Each dose will be administrated intravenously at a constant rate over 30 minutes (500 milliliter per hour [mL/hr]).
  Interventions: Drug: Zanamivir
- Zanamivir 600 mg (Experimental): Subjects will receive a single dose of IV zanamivir 600 mg on Day 1 morning. The repeat dose session will begin on Day 3 evening. Subjects will be receive IV zanamivir 600 mg every 12 hours for 5 days. Each dose will be administrated intravenously at a constant rate over 30 minutes (500 mL/hr).
  Interventions: Drug: Zanamivir

INTERVENTIONS:
Drug: Zanamivir — Zanamivir will be supplied as 10 mg/mL sterile clear, colorless, aqueous solution in 20 mL clear glass vials, each containing 200 mg zanamivir. Intravenous solutions will be prepared with normal saline.

SUMMARY:
Zanamivir is a potent and highly selective inhibitor of the influenza virus neuraminidase. Intravenous (IV) zanamivir is being developed for treatment of hospitalized patients with influenza, especially for those patients who may be in greatest need of parenteral influenza antiviral agents. This study is a pharmacokinetic (PK) study to evaluate the safety/tolerability and pharmacokinetic profiles of IV zanamivir 300 milligrams (mg) and 600 mg in Chinese healthy subjects. Subjects will be randomized to receive either 300 mg or 600 mg IV zanamivir as a single dose followed by repeated dose every 12 hours (h) for 5 days. Subjects will be contacted or will return to study center for a follow-up visit, 7 days after the last dose or withdrawal from the study. Total number of subjects planned for enrollment will be 24 such that approximately 10 subjects complete dosing and critical assessments in each dose cohort. The total duration of the study will be approximately 6 weeks from screening to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination and laboratory tests.
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 19-24 kilogram per meter square (kg/m^2) (inclusive). BMI = (weight in kg)/(height in meters) ^2.
* A female subject is eligible to participate if she is non-childbearing potential or child-bearing potential with negative pregnancy test as determined by urine human chorionic gonadotropin (hCG) test.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in protocol. This criterion must be followed from the time of the first dose of study medication until completion of the follow-up visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Alanine amino transferase (ALT) and bilirubin <=1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Based on single or averaged corrected QT (QTc) values of triplicate ECGs obtained over a brief recording period: QTc <450 milliseconds (msec).

Exclusion Criteria:

* Criteria Based Upon Medical Histories-
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK medical monitor, contraindicates their participation.

Criteria Based Upon Diagnostic Assessments-

* A positive pre-study hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody result within 3 months of screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* A positive test for syphilis.
* Pregnant females as determined by positive urine hCG test at screening or prior to dosing.
* Have a creatinine clearance <=80 milliliter per minute (mL/min) (Cockcroft-Gault).

Estimated creatinine clearance rate (eCCr) = (140 - Age) x Mass (in Kg) x Constant/Serum Creatinine micromole per liter (μmol/L), where constant is 1.23 for men and 1.04 for women.

Other Criteria-

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to the first dosing day in the current study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2015-06-19 (Actual); Study Completion 2015-06-19 (Actual)

PRIMARY OUTCOMES:
Composite of PK parameters of zanamivir following single dose administration | Day 1: Pre-dose and 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 10 h, 12 h and 24 h post-dose
  PK parameter assessed following single dose administration include the observed maximum serum drug concentration (Cmax), time to reach Cmax (tmax), elimination half-time (t1/2), area under the concentration-time curve from administration extrapolated to the last time of quantifiable concentration (AUC [0-t]), area under the concentration-time curve from administration extrapolated to 12 hours of quantifiable concentration (AUC [0-12]), area under the concentration-time curve from time zero extrapolated to infinite time (AUC [0-infinity]), clearance (CL) and volume of distribution after intravenous administration (Vz).
Composite of PK parameters of zanamivir following repeat dose administration | Day 8: Pre-dose and 0.25 h, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 10 h, 12 h and 24 h post-dose
  PK parameter assessed following repeat dose administration include Cmax, pre-dose trough concentration (Ctau), tmax, t1/2, AUC (0-t), area under the concentration-time curve during steady state (AUC [0-tau]), CL, Vz, volume of distribution after intravenous administration at steady state (Vss), observed accumulation ratios (Ro) and time invariance ratio (Rs).

SECONDARY OUTCOMES:
Safety as assessed by the number of subjects with adverse events (AEs) | Up to Day 15
  AEs will be collected from the start of study treatment and until the follow-up contact.
Composite of clinical laboratory assessments as a measure of safety | Up to Day 9
  Absolute values and change over time from pre-dose values of hematology and clinical chemistry parameters will be assessed
Absolute values and change over time from pre-dose values of blood pressure as a measure of safety | Up to Day 9
Absolute values and change over time from pre-dose values of pulse rate as a measure of safety | Up to Day 9
Absolute values and change over time from pre-dose values of respiratory rate as a measure of safety | Up to Day 9
Absolute values and change over time from pre-dose values of temperature as a safety measure | Up to Day 9
Absolute values and change over time from pre-dose values of electrocardiogram (ECG) parameters | Up to Day 9
  A 12-lead ECG will be obtained at each time point during the study and will be evaluated for safety by a qualified physician.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

REFERENCES:
- See also: Results for study 117104 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117104?search=study&b'study_ids=117104'#rs